CLINICAL TRIAL: NCT06619587
Title: A Phase I/II Dose-Escalation and Expansion Study Evaluating the Safety, Pharmacokinetics, and Activity of GDC-7035 as a Single Agent and in Combination With Other Anti-Cancer Therapies in Patients With Advanced Solid Tumors With a KRAS G12D Mutation
Brief Title: A Study to Evaluate Safety, Pharmacokinetics, and Activity of GDC-7035 as a Single Agent and in Combination in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO45416
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I Arm A (Experimental): Dose escalation and expansion arm
  Interventions: Drug: Phase I Arm A
- Phase I Arm B (Experimental): Dose escalation and expansion arm
  Interventions: Drug: Phase I Arm B

INTERVENTIONS:
Drug: Phase I Arm A — Dose escalation and expansion arm, with protocol-defined dose(s) of GDC-7035
  Arms: Phase I Arm A
Drug: Phase I Arm B — Dose escalation and expansion arm, with protocol-defined dose(s) of GDC-7035 in combination with other anti-cancer therapies
  Arms: Phase I Arm B

SUMMARY:
This is a first-in-human Phase I/II, open-label, multicenter, dose-escalation and expansion study designed to evaluate the safety, pharmacokinetics, and preliminary activity of GDC-7035 as a single agent and in combination with other anti-cancer therapies in participants with advanced or metastatic solid tumors that harbor the KRAS G12D mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented advanced or metastatic solid tumor with KRAS G12D mutation
* Agreement to adhere to the contraception requirements described in the protocol for participants of childbearing potential and participants who produce sperm

Exclusion criteria:

* Malabsorption or other condition that would interfere with enteral absorption
* Active brain metastases
* Clinically significant cardiovascular dysfunction or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events, with Severity Determined According to the CTCAE v5.0 Grading Scale | 4 Years
Percentage of Participants with Dose Limiting Toxicity | 4 Years

SECONDARY OUTCOMES:
Plasma Concentrations of GDC-7035 at Specified Timepoints | 4 Years
Blood Concentrations of GDC-7035 at Specified Timepoints | 4 Years
Plasma Concentrations at Specified Timepoints of GDC-7035 Administered in the Fasted State or with a Standardized High-Fat Meal | 4 Years
Blood Concentrations at Specified Timepoints of GDC-7035 Administered in the Fasted State or with a Standardized High-Fat Meal | 4 Years
Objective Response Rate Among Participants | 4 Years
Duration of Response Among Participants | 4 Years
Median Progression Free Survival Time Among Participants | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (36):
- United States (11):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialist-Lake Mary, Lake Mary, Florida
  - University of Illinois, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - START - Midwest - EDOS, Grand Rapids, Michigan
  - Montefiore Einstein Cancer Center, The Bronx, New York
  - Mary Crowley Medical Research Center, Dallas, Pennsylvania
  - Abramson Cancer Center;Univ of Pennsylvania, Philadelphia, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
- Australia (2):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Peter Maccallum Cancer Centre, Parkville, Victoria
- Canada (3):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sir Mortimer B Davis Jewish General Hospital, Montreal, Quebec
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center., Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (6):
  - Instituto de Investigacion Oncologica Vall dHebron (VHIO) - EPON, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - START Madrid_Hospital Universitario HM Sanchinarro_CIOCC, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (4):
  - Western General Hospital;Edinburgh Cancer Center, Edinburgh, Midlothian
  - NIHR UCLH Clinical Research Facility, London
  - The Christie, Manchester
  - Royal Marsden Hospital - Surrey, Sutton

IPD SHARING:
Plan to Share IPD: No